CLINICAL TRIAL: NCT06907056
Title: Effectiveness, Safety, and Tolerability of Darunavir/Cobicistat Plus Lamivudine Versus Darunavir/Cobicistat Plus Tenofovir/Emtricitabine in Virologically Suppressed HIV-1-positive Individuals: 48-week Follow-up in Mexico
Brief Title: Effectiveness and Safety of Darunavir/Cobicistat Plus Lamivudine Versus Darunavir/Cobicistat Plus Tenofovir/Emtricitabine in Virologically Suppressed HIV-1-positive Individuals in Mexico
Acronym: TLALOC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: José Antonio Mata Marín (Other Government)
Responsible Party: Sponsor-Investigator, José Antonio Mata Marín, Doctor, Instituto Mexicano del Seguro Social
Organization: Instituto Mexicano del Seguro Social (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2024-3502-116; R-2024-3502-116 (Other: Instituto Mexicano Del Seguro Social)
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: HIV Infection
Keywords: HIV; dual therapy; DRV/c+3TC; effectiveness; non-inferiority
MeSH Terms: conditions — HIV Infections | interventions — Dual Anti-Platelet Therapy

STUDY DESIGN:
Intervention Model Description: Unicenter, open-label, randomized, noninferiority trial, Participants were randomized to either continue standard therapy or switch to DRV/c+3TC. The primary end point was the proportion of subjects with HIV-1 RNA levels >50 copies/ml after 48 weeks of follow-up, non-inferiority margin of up to 10%. For statistical analysis, data distribution will be identified using the Kolmogorov-Smirnov test; categorical data will be analyzed using the X2 or Fisher test, as appropriate, and will be expressed as numbers and percentages. Quantitative data will be expressed as medians and interquartile ranges or means with standard deviations. A first analysis will be performed at 24 weeks, with follow-up at 48 weeks. The Student's t-test or the Mann-Whitney U-test will be used for data from independent groups according to their distribution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standar therapy (Active Comparator): Darunavir/cobicistat 800/150 mg + tenofovir/emtricitabin 300/200 mg This arm is the commonly used therapy or standard 3-drug therapy consisting of Darunavir/cobicistad 800/150 mg, plus tenofovir/emtricitabine 300/200 mg
  Interventions: Drug: Standard Medical Therapy
- Dual therapy (Experimental): Darunavir/cobicistat 800/150 mg + lamivudine 300 mg This arm is the experimental one, with dual therapy, 2 drugs: darunavir/cobicistat 800/150 mg plus lamivudine 300 mg
  Interventions: Drug: dual therapy

INTERVENTIONS:
Drug: dual therapy — Intervention arm will be dual therapy oh DRV/C 800/150 mg + 3TC 300 mg, this will be compared to standar therapy of 3 drugs with: DRV/c 800/150 mg + TDF/FTC 300/200 mg
  Other Names: DRV/c+3TC
  Arms: Dual therapy
Drug: Standard Medical Therapy — DRV/c+TDF/FTC
  Other Names: DRV/c+TDF/FTC
  Arms: Standar therapy

SUMMARY:
Unicenter, open-label, randomized, noninferiority trial included men with HIV-1 RNA levels <50 copies/ml for at least 6 months on antiretroviral therapy with DRV/c + TFV/FTC (standar therapy), aged over 18 years. Participants were randomized to either continue standard therapy or switch to DRV/c+3TC. The primary end point was the proportion of subjects with HIV-1 RNA levels >50 copies/ml after 48 weeks of follow-up according to the snapshot algorithm, with a non-inferiority margin of up to 10%. For statistical analysis, data distribution will be identified using the Kolmogorov-Smirnov test; categorical data will be analyzed using the X2 or Fisher test, as appropriate, and will be expressed as numbers and percentages. Quantitative data will be expressed as medians and interquartile ranges or means with standard deviations. A first analysis will be performed at 24 weeks, with follow-up at 48 weeks. The Student's t-test or the Mann-Whitney U-test will be used for data from independent groups according to their distribution.

DETAILED DESCRIPTION:
Unicenter, open-label, randomized, noninferiority trial included men with HIV-1 RNA levels <50 copies/ml for at least 6 months on antiretroviral therapy with DRV/c + TFV/FTC (standar therapy), aged over 18 years. Participants were randomized to either continue standard therapy or switch to DRV/c+3TC. The primary end point was the proportion of subjects with HIV-1 RNA levels >50 copies/ml after 48 weeks of follow-up according to the snapshot algorithm, with a non-inferiority margin of up to 10%. For statistical analysis, data distribution will be identified using the Kolmogorov-Smirnov test; categorical data will be analyzed using the X2 or Fisher test, as appropriate, and will be expressed as numbers and percentages. Quantitative data will be expressed as medians and interquartile ranges or means with standard deviations. A first analysis will be performed at 24 weeks, with follow-up at 48 weeks. The Student's t-test or the Mann-Whitney U-test will be used for data from independent groups according to their distribution.

Subject to prior approval of the protocol by the local scientific research ethics committee and the relevant agencies, patients being monitored at the HIV clinic at the Infectious Diseases Hospital of the CMN "La Raza" who are living with HIV and receiving treatment with DRV/c + TFV/FTC for virological suppression will be identified as candidates for participation in the study.

They will be invited to participate in the study protocol, and the project and its likely outcomes will be explained in detail to the subjects. It will be explained that treatment assignment will be randomized using the digital system (MEDSHARING: randomizer for clinical trials) to one of two arms:

1. DRV/c (800 mg/150 mg once daily) + 3TC (300 mg once daily) or
2. DRV/c (800 mg/150 mg once daily) + TFV/FTC (300 mg/200 mg once daily). Answers will be obtained during the medical interview, allowing the patient to freely decide whether to continue or withdraw from the study during the study period without affecting their medical care at the HIV clinic. Informed consent will be obtained, and to maintain privacy, a patient ID number will be assigned at the time of recruitment. Weight (kg), height (cm), body mass index (BMI) (kg/height (m2), body composition (fat, water, muscle, kg, bone, kg) will be measured using the FitScan BC-545F segmental body composition monitor, and waist and hip measurements will be measured using a tape measure. Laboratory studies will include a complete blood count, complete blood chemistry with glucose and creatinine, a complete lipid profile, and post-randomization liver function tests at 4 weeks, 12 weeks, 24 weeks, and 48 weeks post-switch. CD4+ and HIV-1 RNA determinations will be performed prior to randomization, and at 3 months, 6 months, and 12 months post-study entry. Comparisons will be made between measurements taken prior to entry, 24 weeks, and 48 weeks post-study entry. Serum electrolytes (phosphorus, magnesium, calcium), cystatin C, and urinary electrolytes (phosphorus, magnesium, calcium, creatinine, urea, microproteins) will be measured prior to randomization and at 24 and 48 weeks post-switch.

If patients present with elevated AST and/or ALT >90 IU/L, serology tests will be ordered to rule out HBV and HCV.

The ISI, PHQ-9, HADS-A, and HADS-D questionnaires will be administered to assess anxiety, depression, and sleep quality. Additionally, the HIVTSQ questionnaire will be administered to assess treatment satisfaction at weeks 4, 12, 24, and 48 weeks post-randomization, and the HIV-SDM questionnaire will be administered to assess HIV-related symptoms and distress. At each medical visit, potential drug-related adverse effects will be deliberately inquired about by device and system, and will be classified into four grades using the DAIDS adverse event scale.

ELIGIBILITY:
Inclusion Criteria:

* Men with HIV infection who are virologically suppressed with DRV/c (800 mg/150 mg) + TFV/FTC (300 mg/200 mg) for at least 6 months
* Age ≥18 years-70 years
* eGFR ≥30 mL/min
* Written informed consent
* Beneficiaries of the Mexican Social Security Institute treated at the Infectious Diseases Hospital of the La Raza National Medical Center.

Exclusion Criteria:

* Withdrawal of informed consent
* Loss of medical insurance
* Presence of tuberculosis or other opportunistic infection requiring adjustment of the ARV regimen
* Incomplete data collected during visits Uncontrolled chronic gastrointestinal conditions Desire to be on a single-dose regimen Coinfection with hepatitis B virus during follow-up if in the DRV/3TC arm Coinfection with hepatitis C virus during follow-up

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | 48 weeks
  Individuals with >50 copies/ml

SECONDARY OUTCOMES:
Non-inferiority | 48 weeks
  Delta between standard and experimental therapy <10%
Safety | 48 weeks
  Adverse events by group and drug tolerability will be reported by device and system, and their severity will be based on the Division of AIDS (DAIDS) Antiretroviral Drug-Associated Adverse Event Severity Scale, which categorizes them in severity from 1 to 4. Grade 1: Mild or no harm; Grade 2: Moderate adverse events or minimal interference with social and functional activities; Grade 3: Severe symptoms causing inability to perform social/functional activities or requiring hospitalization. Grade IV: Those that are life-threatening with symptoms causing inability to perform basic self-care and where intervention is required to prevent permanent deterioration or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Infectología, Centro Médico Nacional La Raza, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
The data cannot be shared openly because it contains personal information about the participants; if required, it can be requested from the corresponding author.

REFERENCES:
- [Background] Figueroa MI, Sued O, Cecchini D, Sanchez M, Rolon MJ, Lopardo G, Ceschel M, Mernies G, De Stefano M, Patterson P, Gun A, Fink V, Ortiz Z, Cahn P; ANDES Study Group. Dual therapy based on co-formulated darunavir/ritonavir plus lamivudine for initial therapy of HIV infection: The ANDES randomized controlled trial. Int J Antimicrob Agents. 2024 Oct;64(4):107301. doi: 10.1016/j.ijantimicag.2024.107301. Epub 2024 Aug 14. PMID 39151647
- [Background] Pulido F, Ribera E, Lagarde M, Perez-Valero I, Palacios R, Iribarren JA, Payeras A, Domingo P, Sanz J, Cervero M, Curran A, Rodriguez-Gomez FJ, Tellez MJ, Ryan P, Barrufet P, Knobel H, Rivero A, Alejos B, Yllescas M, Arribas JR; DUAL-GESIDA-8014-RIS-EST45 Study Group. Dual Therapy With Darunavir and Ritonavir Plus Lamivudine vs Triple Therapy With Darunavir and Ritonavir Plus Tenofovir Disoproxil Fumarate and Emtricitabine or Abacavir and Lamivudine for Maintenance of Human Immunodeficiency Virus Type 1 Viral Suppression: Randomized, Open-Label, Noninferiority DUAL-GESIDA 8014-RIS-EST45 Trial. Clin Infect Dis. 2017 Nov 29;65(12):2112-2118. doi: 10.1093/cid/cix734. PMID 29020293
- [Background] Fabbiani M, Gagliardini R, Ciccarelli N, Quiros Roldan E, Latini A, d'Ettorre G, Antinori A, Castagna A, Orofino G, Francisci D, Chinello P, Madeddu G, Grima P, Rusconi S, Del Pin B, Lombardi F, D'Avino A, Foca E, Colafigli M, Cauda R, Di Giambenedetto S, De Luca A; ATLAS-M Study Group. Atazanavir/ritonavir with lamivudine as maintenance therapy in virologically suppressed HIV-infected patients: 96 week outcomes of a randomized trial. J Antimicrob Chemother. 2018 Jul 1;73(7):1955-1964. doi: 10.1093/jac/dky123. PMID 29668978
- [Background] Perez-Molina JA, Rubio R, Rivero A, Pasquau J, Suarez-Lozano I, Riera M, Estebanez M, Santos J, Sanz-Moreno J, Troya J, Marino A, Antela A, Navarro J, Esteban H, Moreno S; GESIDA 7011 Study Group. Dual treatment with atazanavir-ritonavir plus lamivudine versus triple treatment with atazanavir-ritonavir plus two nucleos(t)ides in virologically stable patients with HIV-1 (SALT): 48 week results from a randomised, open-label, non-inferiority trial. Lancet Infect Dis. 2015 Jul;15(7):775-84. doi: 10.1016/S1473-3099(15)00097-3. Epub 2015 Jun 7. Erratum In: Lancet Infect Dis. 2015 Sep;15(9):998. doi: 10.1016/S1473-3099(15)00241-8. PMID 26062881
- [Background] Cahn P, Andrade-Villanueva J, Arribas JR, Gatell JM, Lama JR, Norton M, Patterson P, Sierra Madero J, Sued O, Figueroa MI, Rolon MJ; GARDEL Study Group. Dual therapy with lopinavir and ritonavir plus lamivudine versus triple therapy with lopinavir and ritonavir plus two nucleoside reverse transcriptase inhibitors in antiretroviral-therapy-naive adults with HIV-1 infection: 48 week results of the randomised, open label, non-inferiority GARDEL trial. Lancet Infect Dis. 2014 Jul;14(7):572-80. doi: 10.1016/S1473-3099(14)70736-4. Epub 2014 Apr 27. PMID 24783988
- [Background] Achhra AC, Mwasakifwa G, Amin J, Boyd MA. Efficacy and safety of contemporary dual-drug antiretroviral regimens as first-line treatment or as a simplification strategy: a systematic review and meta-analysis. Lancet HIV. 2016 Aug;3(8):e351-e360. doi: 10.1016/S2352-3018(16)30015-7. Epub 2016 May 31. PMID 27470027
- [Background] Corado KC, Caplan MR, Daar ES. Two-drug regimens for treatment of naive HIV-1 infection and as maintenance therapy. Drug Des Devel Ther. 2018 Nov 1;12:3731-3740. doi: 10.2147/DDDT.S140767. eCollection 2018. PMID 30464404
- [Background] Trujillo-Rodriguez M, Munoz-Muela E, Serna-Gallego A, Milanes-Guisado Y, Praena-Fernandez JM, Alvarez-Rios AI, Herrera-Hidalgo L, Dominguez M, Lozano C, Romero-Vazquez G, Roca C, Espinosa N, Gutierrez-Valencia A, Lopez-Cortes LF. Immunological and inflammatory changes after simplifying to dual therapy in virologically suppressed HIV-infected patients through week 96 in a randomized trial. Clin Microbiol Infect. 2022 Aug;28(8):1151.e9-1151.e16. doi: 10.1016/j.cmi.2022.02.041. Epub 2022 Mar 11. PMID 35289296
- [Background] Consolidated Guidelines on HIV Prevention, Testing, Treatment, Service Delivery and Monitoring: Recommendations for a Public Health Approach [Internet]. Geneva: World Health Organization; 2021 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK572729/ PMID 34370423